CLINICAL TRIAL: NCT04893629
Title: The Effectiveness of Autologous Mono Nuclear Cells in the Treatment of Dilated Cardiomyopathy in Children
Brief Title: New Horizons for the Treatment of Cardiomyopathy in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of necessary equipment
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDMS-Cardio-01-2021
Record Dates: First submitted 2021-03-24; First posted 2021-05-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cardiomyopathy
Keywords: Dilated; Cardio-myopathy; pediatric; mono; nuclear; cells
MeSH Terms: conditions — Cardiomyopathies; Dilatation, Pathologic | interventions — Furosemide; Captopril

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): children diagnosed with dilated cardiomyopathy , will undergo trans endocardium injection of mono nuclear cells
  Interventions: Biological: mono nuclear cells injection
- control group (Active Comparator): children diagnosed with dilated cardiomyopathy ,will continue the classic medical treatment
  Interventions: Drug: Digoxin+furosemide+captopril

INTERVENTIONS:
Biological: mono nuclear cells injection — trans endocardium injection of autologous mono nuclear cells for the intervention group and classic treatment for the control group
  Arms: intervention group
Drug: Digoxin+furosemide+captopril — classical heart failure medical treatment
  Other Names: lasix,capoten
  Arms: control group

SUMMARY:
Collecting mono nuclear cells from the patient's blood after a course of granulocyte stimulation then injecting them into the weak heart muscle measuring the heart function at the beginning and after 2.4.6 months to assess the improvement due to this procedure, by comparing these patients to patients with the same condition treated the classic way.

DETAILED DESCRIPTION:
Dilated cardiomyopathy in children has high morbidity and mortality, current treatment doesn't improve the prognosis and the only cure available is heart transplantation which is limited, has long waiting list (if available), high cost, and has many side effects, leading to the need of novel effective, less costly therapeutic alternatives.

Stem cell therapy has proven to improve the cardiac function, reverse the pathologic histological changes, decrease the morbidity and mortality, offering a possible replacement to heart transplantation, different reports proved the safety and efficacy of this therapy using different types of cells and different routs of application in cardiomyopathy and acute myocardial infarction in children and adults, and in congenital heart disease, but the published cases of this therapy conducted on children with dilated cardiomyopathy are scanty .

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy diagnosed and treated at least 6 mo. Ago
* LVEF less than 40%
* Use of I.V inotropes

Exclusion Criteria:

* Acute infection
* Severe organ failure (other than the heart)

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Left ventricle ejection fraction (LVEF) | 6 months
  measured by echo (mono mode, 3 Dimentional)

CONTACTS AND LOCATIONS:
Overall Officials: samir srour, prof, Study Chair — membership of the French society of the pediatric cardiology
Locations (1):
- Children'S Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selem SM, Kaushal S, Hare JM. Stem cell therapy for pediatric dilated cardiomyopathy. Curr Cardiol Rep. 2013 Jun;15(6):369. doi: 10.1007/s11886-013-0369-z. PMID 23666883
- [Background] Zeinaloo A, Zanjani KS, Bagheri MM, Mohyeddin-Bonab M, Monajemzadeh M, Arjmandnia MH. Intracoronary administration of autologous mesenchymal stem cells in a critically ill patient with dilated cardiomyopathy. Pediatr Transplant. 2011 Dec;15(8):E183-6. doi: 10.1111/j.1399-3046.2010.01366.x. Epub 2010 Sep 29. PMID 20880092
- [Background] Vrtovec B, Poglajen G, Lezaic L, Sever M, Domanovic D, Cernelc P, Socan A, Schrepfer S, Torre-Amione G, Haddad F, Wu JC. Effects of intracoronary CD34+ stem cell transplantation in nonischemic dilated cardiomyopathy patients: 5-year follow-up. Circ Res. 2013 Jan 4;112(1):165-73. doi: 10.1161/CIRCRESAHA.112.276519. Epub 2012 Oct 12. PMID 23065358
- [Background] Abdel-Latif A, Bolli R, Tleyjeh IM, Montori VM, Perin EC, Hornung CA, Zuba-Surma EK, Al-Mallah M, Dawn B. Adult bone marrow-derived cells for cardiac repair: a systematic review and meta-analysis. Arch Intern Med. 2007 May 28;167(10):989-97. doi: 10.1001/archinte.167.10.989. PMID 17533201
- [Background] Mozid AM, Arnous S, Sammut EC, Mathur A. Stem cell therapy for heart diseases. Br Med Bull. 2011;98:143-59. doi: 10.1093/bmb/ldr014. Epub 2011 May 19. PMID 21596713
- See also: -Wang et al. Stem Cell Research & Therapy (2019) 10:137 — https://doi.org/10.1186/s13287-019-1238-5
- See also: I. M-Behnke et al. Regenerative therapies in young hearts with structural or congenital heart disease — http://dx.doi.org/10.21037/tp.2019.03.01